CLINICAL TRIAL: NCT07269626
Title: A Prospective Phase II Study of Systemic Therapy With Combined Personalized Ultrafractionated Stereotactic Adaptive Radiation Therapy (PULSAR) in Pancreatic Cancer
Brief Title: PULSAR in Systemic Therapy for Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARIS-PC; 2025-09-076 (Other: Samsung Medical Center IRB)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma; Borderline Resectable Pancreatic Ductal Adenocarcinoma; Oligometastatic Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic cancer; proton beam radiotherapy; PULSAR
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Standard systemic therapy with PULSAR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PULSAR (Experimental): Standard systemic therapy with PULSAR
  Interventions: Radiation: Personalized Ultrafractionated Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Personalized Ultrafractionated Adaptive Radiotherapy — Proton therapy will be delivered at 12 gray (relative biological effectiveness, RBE) per fraction, administered once every 3 to 4 weeks, for a total of 2 to 3 fractions.

SUMMARY:
Pancreatic cancer remains one of the malignancies with the lowest survival rates, largely due to late-stage diagnosis and the difficulty of achieving curative resection. A substantial proportion of patients present with locally advanced, unresectable disease at the time of diagnosis, making intensive systemic therapy the current standard of care. For selected patients, radiation therapy (RT) is integrated to improve local control. Local progression in the pancreas can lead to severe complications, including intractable pain, gastric outlet obstruction, and biliary obstruction, which ultimately contribute to morbidity, deteriorating quality of life, and reduced overall survival. Therefore, effective local therapy remains a critical component of comprehensive management.

However, delivering high-dose radiation to pancreatic tumors is particularly challenging because the pancreas is anatomically surrounded by radiation-sensitive organs such as the stomach, duodenum, liver, kidneys, and small bowel. Conventional RT and stereotactic body RT (SBRT) have both been limited by gastrointestinal toxicity, making substantial dose escalation difficult and resulting in modest local control outcomes.

Previous studies combining systemic therapy with radiotherapy have shown signals of improved local progression-free survival (LPFS) and progression-free survival (PFS). Still, results have been inconsistent across trials, highlighting the need for rigorous clinical evaluation of the true therapeutic benefit of integrating radiotherapy with systemic treatment in this disease population.

Conventional RT often requires several weeks of treatment, during which interruption or modification of systemic therapy may increase the risk of distant progression. SBRT shortens the treatment duration but exposes patients to large per-fraction radiation doses, increasing the risk of gastrointestinal injury and limiting eligibility to highly selected cases.

Against this backdrop, the recently proposed PULSAR (Personalized Ultra-fractionated Stereotactic Adaptive Radiotherapy) strategy offers an innovative approach to overcome the limitations of traditional radiation therapy. PULSAR delivers 3-4 ultra-fractionated, stereotactic "pulses" of radiation at intervals of approximately 3-4 weeks. Each pulse is delivered with adaptive planning based on interval changes in tumor anatomy and nearby organs at risk. This wide spacing minimizes interruptions to systemic therapy and provides time for tumor shrinkage and normal tissue recovery before subsequent pulses. These features may reduce toxicity while enabling more effective dose delivery to the tumor. Such advantages are particularly relevant for pancreatic tumors located adjacent to sensitive gastrointestinal structures, potentially improving upon the limitations of SBRT.

The proton beam therapy offers additional precision through the physical characteristics of proton beams, particularly the Bragg peak, which allows for high-dose deposition within the tumor while sparing surrounding normal tissues. The combination of proton therapy with the PULSAR framework may provide a highly targeted, organ-preserving local treatment strategy for a disease known for its complex anatomy and therapeutic difficulty.

Within this context, a clinical strategy that integrates intensive first-line systemic therapy followed by PULSAR-based adaptive proton radiotherapy holds promising potential. Systemic therapy may reduce tumor burden, after which personalized, pulse-based proton irradiation can be tailored according to treatment response, delivering biologically effective doses to maximize local control while maintaining systemic treatment intensity. This approach may enhance survival outcomes by addressing both local disease control and risk of distant metastasis.

In summary, given the critical need to improve survival in locally advanced pancreatic cancer and the inherent limitations of existing radiation approaches, combining PULSAR-guided adaptive proton therapy with contemporary systemic therapy represents a compelling new treatment paradigm. This study aims to systematically evaluate the clinical feasibility, safety, and therapeutic effectiveness of this integrated approach in patients with locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Histologically confirmed pancreatic ductal adenocarcinoma.
* Disease extent classified as borderline resectable, locally advanced, or oligometastatic disease (defined as ≤ 3 metastatic lesions) at the time of staging evaluation.
* Completion of at least 2-4 cycles of first-line systemic therapy (FOLFIRINOX, gemcitabine/nab-paclitaxel, or NALIRIFOX) without evidence of distant progression.
* Presence of a lesion suitable for radiotherapy, as determined by the investigator, and measurable disease per RECIST 1.1 criteria.
* Ability to understand the study requirements and voluntarily provide written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Presence of brain metastases or leptomeningeal disease.
* History of prior radiotherapy to the intended treatment area.
* Significant comorbid conditions that may interfere with study participation or the ability to safely receive study treatment, as determined by the investigator (e.g., uncontrolled infection, congestive heart failure, clinically significant arrhythmia, or severe psychiatric illness).
* Patients deemed unlikely to comply with study procedures or follow-up requirements.
* Any condition that, in the opinion of the principal investigator or treating physician, makes the patient inappropriate for participation in this trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival at 1-year after enrollment | PFS rate at 1 year is defined as the proportion of patients who have not experienced disease progression or death within 12 months from study enrollment.
  PFS is defined as the period from the date of the first PULSAR session to the date of documented disease progression, death, or last follow-up, whichever occurs first.
Progression-free survival | at 1 year-progression-free survival (PFS_, defined as the proportion of patients who have not experienced disease progression or death within 12 months from study enrollment.
  Defined as the period from the date of the study enrollment to the date of documented disease progression, death, or last follow-up, whichever occurs first.
Local control (LC) | The 2-year LC rate will be defined as the proportion of patients who remain free from local tumor progression at 2 years after study enrollment.
  LC is defined as proportion of patients without local tumor progression based on RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Overall survival | OS rate at 2-year, is defined as the proportion of patients who remain alive at 2 years after study enrollment.
  Overall survival (OS) is defined as the period from the date of the enrollment to the date of documented death, or last follow-up, whichever occurs first.
Objective Response Rate (ORR) | ORR will be assessed according to RECIST version 1.1 at 1 month after completion of PULSAR (with an allowable window of up to 8 weeks).
  ORR will be assessed according to RECIST version 1.1 at 1 month after completion of PULSAR (with an allowable window of up to 8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Il Yu, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Select Province/State, South Korea

IPD SHARING:
Plan to Share IPD: No